CLINICAL TRIAL: NCT02302287
Title: Gut-kidney Axis: Renal Effects of Meditarranean Diet and Low-protein Diet With Ketoacids to Restore Physiological Intestinal Mibrobiota in Chronic Kidney Disease
Brief Title: Renal Effects of Meditarranean Diet and Low-protein Diet With Ketoacids on Physiological Intestinal Mibrobiota in CKD
Acronym: MEDIKA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Sanitaria ASL Avellino 2 (Other)
Responsible Party: Principal Investigator, Dr Biagio Di Iorio, Chair of Nephrology Departement, Azienda Sanitaria ASL Avellino 2
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: rf 2013-02355394
Record Dates: First submitted 2014-11-21; First posted 2014-11-27 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Renal Insufficiency
Keywords: Chronic kidney disease; mediterranean diet; low-protein diet; ketoacids; intestinal microbiota
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): 1. Free diet for 3 months: protein 1 g/body weight/day (animal protein 50-70 g/day, plant protein 15-20 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 1,2-1,5 g/day; sodium 6 g/day, potassium 2-4 g/day;
  2. Ketoacids diet for 6 months: protein 0,3-0,5 g/bw/day (animal protein 0 g/day, plant protein 30-40 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 0,6-0,8 g/day; sodium 6 g/day, potassium 2-4 g/day; mixture of essential aminoacids and ketoacids 0,05 g/kg ideal bw/day
  3. Mediterranean diet for 6 months: protein 0,7-0,8 g/bw/day (animal protein 30-40 g/day, plant protein 40-50 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 1,2-1,5 g/day; sodium 2,5-3 g/day, potassium 2-4 g/day
  4. Mediterranean diet and ketoacids for 6 months
  Interventions: Dietary Supplement: Ketoacids diet; Other: Mediterranean diet; Other: Free diet
- Group B (Experimental): 1. Free diet for 3 months: protein 1 g/body weight/day (animal protein 50-70 g/day, plant protein 15-20 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 1,2-1,5 g/day; sodium 6 g/day, potassium 2-4 g/day;
  2. Mediterranean diet for 6 months: protein 0,7-0,8 g/bw/day (animal protein 30-40 g/day, plant protein 40-50 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 1,2-1,5 g/day; sodium 2,5-3 g/day, potassium 2-4 g/day;
  3. Ketoacids diet for 6 months: protein 0,3-0,5 g/bw/day (animal protein 0 g/day, plant protein 30-40 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 0,6-0,8 g/day; sodium 6 g/day, potassium 2-4 g/day; mixture of essential aminoacids and ketoacids 0,05 g/kg ideal bw/day
  4. Mediterranean diet and ketoacids for 6 months
  Interventions: Dietary Supplement: Ketoacids diet; Other: Mediterranean diet; Other: Free diet
- Group control (Other): Free diet: protein 1 g/body weight/day (animal protein 50-70 g/day, plant protein 15-20 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 1,2-1,5 g/day; sodium 6 g/day, potassium 2-4 g/day
  Interventions: Other: Free diet

INTERVENTIONS:
Dietary Supplement: Ketoacids diet — Ketoacids diet for 6 months: protein 0,3-0,5 g/bw/day (animal protein 0 g/day, plant protein 30-40 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 0,6-0,8 g/day; sodium 6 g/day, potassium 2-4 g/day; mixture of essential aminoacids and ketoacids 0,05 g/kg ideal bw/day
  Other Names: KD
  Arms: Group A; Group B
Other: Mediterranean diet — Mediterranean diet for 6 months: protein 0,7-0,8 g/bw/day (animal protein 30-40 g/day, plant protein 40-50 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 1,2-1,5 g/day; sodium 2,5-3 g/day, potassium 2-4 g/day
  Other Names: MD
  Arms: Group A; Group B
Other: Free diet — Free diet for 3 months: protein 1 g/body weight/day (animal protein 50-70 g/day, plant protein 15-20 g/day); energy 30-35 kcal/bw/day; Calcium 1,1-1,3 g, phosphate 1,2-1,5 g/day; sodium 6 g/day, potassium 2-4 g/day;
  Other Names: FD

SUMMARY:
Food intake has a deep influence on gut microbiota composition and function, both in health and in disease status. In chronic kidney disease (CKD), a microbiota dysbiosis status is observed. Moreover, many toxic uremic molecules are microbial-derived and their accumulation promotes, in turn, disease progression.

Investigators' hypothesis foresees a beneficial effect of nutritional treatments, able to restore gut microbiota balance, to lower microbial-derived uremic toxins and to improve clinical conditions in CKD patients.

Mediterranean Diet (MD) is supposed to have beneficial effect on microbiota composition, while low-protein diet supplemented with ketoacids (KD) is used in CKD patients for the improvement of clinical conditions, but its effects on gut microbiota are currently unknown. Investigators' project aim is to verify the effects of MD and KD on: microbiota and metabolome composition, microbial-derived uremic toxins level and clinical conditions in a cohort of CKD patients.

DETAILED DESCRIPTION:
Background: In CKD the biochemical milieu of gastrointestinal tract (GI) is altered by several mechanisms, affecting gut microbiota composition and function. Beyond exerting metabolic functions, microbiota influences the general healthy status. It digests food mainly through saccharolytic or proteolytic catabolism, with a prevalence of the former in healthy status. On the contrary, in CKD, dysbiosis with the prevalence of the latter is observed.

In this setting, reduction in glomerular filtration rate and increase in urea levels result in its heavy influx into the GI. Here urea is hydrolyzed spontaneously and/or by microbial urease, releasing ammonia, readily converted into ammonium hydroxide. The latter raises GI pH, causing mucosa irritation, enterocolitis and changes in microbiota composition. This contributes to worsening of inflammation and disease progression: indeed, microbiota has been identified as the primary source of several well known and yet unidentified volatile organic compounds (VOC), including some of the main uremic toxins.

Some beneficial effects observed from studies with low-protein diet supplemented with ketoacids in CKD cannot be solely explained by the reduced protein intake. Investigators' hypothesis is that ketoacids may have direct protective effects on renal damage progression, through induced modifications in gut biochemical milieu and in microbiota composition.

Similarly, the Mediterranean Diet with its fibers supply can contribute to restore gut microbiota balance.

Hypothesis:

The first hypothesis foresees a beneficial effect of KD on microbiota balancing and microbial-derived uremic toxins decrease in CKD patients, through KD-induced urea reduction. The second envisages MD direct effects on gut microbiota composition with an increase in protective species and a decrease in uremic toxins production.

The study will evaluate the effects of three different dietary regimens, composed as follows:

FD contains 1 g/bw/day of protein, plant protein 15-20 g/day;

* MD contains 0.7-0.8 g/bw/day of protein, plant protein 40-50 g/day;
* KD contains 0.3-0.5 g/bw/day of protein, animal protein zero g/day, plant protein 30-40 g/day, plus ketoacids of 0.05 g/bw/day.

Specific aim:

1. To evaluate the effects of Mediterranean diet (MD) and low-protein diet supplemented with ketoacids (KD) on microbiota composition
2. To evaluate the effects of KD and MD on microbial-derived VOC (already identified and yet unidentified uremic toxins) levels by metabolomics
3. To evaluate the effects of KD or MD on renal function parameters, uremia, inflammatory and nutritional status

Experimental Design Aim 1:

The designed study will be experimental, randomized, cross-over. It will be carried out according to the Declaration of Helsinki (IV Adaptation) and will be submitted to the approval of the local Ethics Committee; written consent will be obtained from all subjects. 60 patients with CKD stages 3b-4 (MDRD formula) will be enrolled, according to the inclusion and exclusion criteria (see below).

Experimental Design Aim 2:

Untarget metabolomic analysis will be carried out on fecal and urine samples collected at the same time points described in Experimental design aim 1 for VOC (GC-MS/MS) and non-VOC profiling (LC-MS/MS). Sera collected at the same time points will be also analyzed by untarget metabolomic for non-VOC profiling and by target metabolomic to quantify the already known uremic toxins, namely indoxyl sulfate and p-cresyl sulfate, and potential metabolite biomarkers found by the untarget experiment.

Experimental Design Aim 3:

Additionally, each patient will undergo medical examination every three months, with evaluation of: blood pressure and nutritional status. Moreover, at the same time points of aim 1 (T0, T3, T9, T12 and T18 months from the beginning of the study) each patient will provide blood and urine samples, both for routine and experimental analysis.

ELIGIBILITY:
Inclusion Criteria:

* prevalent patients in tertiary nephrology clinic;
* patients over 18 years;
* CKD stage 3b-4 (eGFR between 15 and 45 ml/min/1.73m2, estimated by MDRD formula);
* clinically proven adherence to prescribed therapies;
* informed consent signed.

Exclusion Criteria:

* change of GFR >30% within the last 3 months;
* acute, intercurrent disease during the previous 3 months;
* severe undernutrition as indicated by: BMI < 20 kg/m2 and serum albumin < 3.2 g/dl, or BMI < 17.5 kg/m2 whatever albumin value, or body weight reduction > 5% within the last month or > 10% within the last six months;
* pregnancy or feeding;
* chronic treatment with steroid or cytotoxic drugs; fast progressing glomerulonephritis; active SLE and vasculitis;
* gastrointestinal diseases (Crohn disease, Ulcerative colitis, Celiac Sprue, Stypsis); 7) infectious diseases; 8) cardiac failure stage III-IV NYHA; advanced liver cirrhosis; active cancer diseases; severe encephalopathy associated with lack of spontaneous feeding; chronic obstructive respiratory diseases needing oxygen treatment; 9) use of antibiotics or probiotics until 15 days before the enrolment; 10) psychiatric disease or inability to assess follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in fecal microbiota by MD and KD at 18 months | 0-18 months from the beginning of the study
  Active fecal microbiota will be analyzed a culture-independent methods. Bacterial tag encoded FLX-titanium amplican pyrosequencing (bTEFAP) analyses will be carried out for bacterial RNA directly extracted from feces at months 0, 3, 9, 12 and 18.

SECONDARY OUTCOMES:
Change from baseline in microbial-derived uremic toxins level at 18 months | 0-18 months from the beginning of the study
  Untarget metabolomic analysis will be carried out on fecal and urine samples collected at months 0,3,9,12 and 18 after the beginning of the study for volatile organic compounds (VOC) (GC-MS/MS) and non-VOC profiling (LC-MS/MS). Sera collected at the same time points will be also analyzed by untarget metabolomic for non-VOC profiling and by target matabolomic to quantify uremic toxins, as indoxyl sulfate and p-cresyl sulfate, and potential metabolite biomarkers found by the untarget experiment
Change from baseline in renal function at 18 months | 0-18 months from the beginning of the study
  each patient will provide at months 0,3,9,12 and 18 blood and urine samples for routine analyses to measure urea, creatinine, estimated glomerular filtration rate, BUN, blood pressure, proteinuria
Change from baseline in nutritional status at 18 months | 0-18 months from the beginning of the study
  each patient will provide at months 0,3,9,12 and 18 blood and urine samples for routine analyses to measure acid-basic balance, serum and urine electrolytes, PTH, serum proteins, haemoglobin,
Change from baseline in inflammatory status at 18 months | 0-18 months from the beginning of the study
  each patient will provide at months 0,3,9,12 and 18 blood and urine samples for routine analyses to measure EGF/MCP-1 ratio, CRP, TNF-a, IL-6
Change from baseline in microbial-derived uremic toxins level at 18 months | 0-18 months from the beginning of the study
  Sera will be collected at months 0,3,9,12 and 18 after the beginning of the study to quantify uremic toxin Cyanate

CONTACTS AND LOCATIONS:
Overall Officials: Biagio Raffaele Di Iorio, PI, Principal Investigator — Azienda Sanitaria ASL Avellino 2
Locations (1):
- UOC Nefrologia, Solofra, Avellino, Italy

REFERENCES:
- [Background] Bellizzi V, Chiodini P, Cupisti A, Viola BF, Pezzotta M, De Nicola L, Minutolo R, Barsotti G, Piccoli GB, Di Iorio B. Very low-protein diet plus ketoacids in chronic kidney disease and risk of death during end-stage renal disease: a historical cohort controlled study. Nephrol Dial Transplant. 2015 Jan;30(1):71-7. doi: 10.1093/ndt/gfu251. Epub 2014 Jul 30. PMID 25082793
- [Background] Bellizzi V, Di Iorio BR, De Nicola L, Minutolo R, Zamboli P, Trucillo P, Catapano F, Cristofano C, Scalfi L, Conte G; ERIKA Study-group. Very low protein diet supplemented with ketoanalogs improves blood pressure control in chronic kidney disease. Kidney Int. 2007 Feb;71(3):245-51. doi: 10.1038/sj.ki.5001955. Epub 2006 Oct 11. PMID 17035939
- [Background] Marzocco S, Dal Piaz F, Di Micco L, Torraca S, Sirico ML, Tartaglia D, Autore G, Di Iorio B. Very low protein diet reduces indoxyl sulfate levels in chronic kidney disease. Blood Purif. 2013;35(1-3):196-201. doi: 10.1159/000346628. Epub 2013 Mar 13. PMID 23485887
- [Background] Di Iorio BR, Bellizzi V, Bellasi A, Torraca S, D'Arrigo G, Tripepi G, Zoccali C. Phosphate attenuates the anti-proteinuric effect of very low-protein diet in CKD patients. Nephrol Dial Transplant. 2013 Mar;28(3):632-40. doi: 10.1093/ndt/gfs477. Epub 2012 Nov 19. PMID 23166309
- [Background] Di Iorio BR, Minutolo R, De Nicola L, Bellizzi V, Catapano F, Iodice C, Rubino R, Conte G. Supplemented very low protein diet ameliorates responsiveness to erythropoietin in chronic renal failure. Kidney Int. 2003 Nov;64(5):1822-8. doi: 10.1046/j.1523-1755.2003.00282.x. PMID 14531817
- [Background] De Angelis M, Montemurno E, Piccolo M, Vannini L, Lauriero G, Maranzano V, Gozzi G, Serrazanetti D, Dalfino G, Gobbetti M, Gesualdo L. Microbiota and metabolome associated with immunoglobulin A nephropathy (IgAN). PLoS One. 2014 Jun 12;9(6):e99006. doi: 10.1371/journal.pone.0099006. eCollection 2014. PMID 24922509
- [Background] Scalone L, Borghetti F, Brunori G, Viola BF, Brancati B, Sottini L, Mantovani LG, Cancarini G. Cost-benefit analysis of supplemented very low-protein diet versus dialysis in elderly CKD5 patients. Nephrol Dial Transplant. 2010 Mar;25(3):907-13. doi: 10.1093/ndt/gfp572. Epub 2009 Dec 14. PMID 20008828
- [Background] Brunori G, Viola BF, Parrinello G, De Biase V, Como G, Franco V, Garibotto G, Zubani R, Cancarini GC. Efficacy and safety of a very-low-protein diet when postponing dialysis in the elderly: a prospective randomized multicenter controlled study. Am J Kidney Dis. 2007 May;49(5):569-80. doi: 10.1053/j.ajkd.2007.02.278. PMID 17472838